CLINICAL TRIAL: NCT01864317
Title: Assessment of Optic Nerve Radiation in Patients With Glaucoma and Ocular Hypertension by 7 Tesla Diffusion Tensor Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-220213
Record Dates: First submitted 2013-05-03; First posted 2013-05-29 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension; Normal Tension Glaucoma
Keywords: 7-Tesla Magnetic Resonance Imaging; Intraocular Pressure; Retinal Nerve Fiber Thickness; Visual Field Test
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Low Tension Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Primary Open Angle Glaucoma (Experimental): 30 patients with primary open angle glaucoma
  Interventions: Device: 7-Tesla MRI; Other: Optical Coherence Tomography; Other: Heidelberg Retina Tomography; Other: Scanning Laser Polarimetry; Other: Humphrey Perimetry; Other: Applanation Tonometry
- Normal Tension Glaucoma (Experimental): 30 patients with normal tension glaucoma
  Interventions: Device: 7-Tesla MRI; Other: Optical Coherence Tomography; Other: Heidelberg Retina Tomography; Other: Scanning Laser Polarimetry; Other: Humphrey Perimetry; Other: Applanation Tonometry
- Ocular Hypertension (Experimental): 30 patients with ocular hypertension
  Interventions: Device: 7-Tesla MRI; Other: Optical Coherence Tomography; Other: Heidelberg Retina Tomography; Other: Scanning Laser Polarimetry; Other: Humphrey Perimetry; Other: Applanation Tonometry
- Healthy subjects (Other): 30 healthy control subjects
  Interventions: Device: 7-Tesla MRI; Other: Optical Coherence Tomography; Other: Heidelberg Retina Tomography; Other: Scanning Laser Polarimetry; Other: Humphrey Perimetry; Other: Applanation Tonometry

INTERVENTIONS:
Device: 7-Tesla MRI — High resolution functional and structural imaging of the visual pathway
Other: Optical Coherence Tomography — Measurement of retinal nerve fiber thickness
Other: Heidelberg Retina Tomography — Measurement of retinal nerve fiber thickness
Other: Scanning Laser Polarimetry — Measurement of retinal nerve fiber thickness
Other: Humphrey Perimetry — Visual Field Testing
Other: Applanation Tonometry — Measurement of Intraocular Pressure

SUMMARY:
Glaucoma is among the leading causes for blindness in the western world. Elevated intraocular pressure (IOP) has been identified as the most important risk factor. However, some patients progress despite adequate IOP lowering while some subjects with elevated IOP never develop glaucoma. Other patients develop glaucoma although IOP measurements were always in the normal range. Therefore, other factors must be involved. In the last years, studies using MRI have been performed and evidence has accumulated that also changes in retrobulbar structures are present, in particular in the lateral geniculate nucleus and the visual cortex. However, these studies were limited by the low spatial resolution of the MRI instruments used.

The investigators propose to overcome this problem by using an ultrahigh-field Magnetom 7T whole-body MR scanner (Siemens Medical, Germany) installed at the MR Centre of Excellence at the Medical University of Vienna. This scanner is equipped with a 32-channel head coil and the SC72 high-performance gradient system and is thus perfectly suited for structural and functional imaging. The aim of the present study is to investigate whether structural and functional parameters are altered in patients with primary open angle glaucoma (POAG), normal tension glaucoma (NTG), ocular hypertension (OHT) compared to healthy control subjects. The exact topographical survey of intracranial structures such as the LGN and the assessment of neuronal structures by DTI may allow for the better assessment of therapeutic responses to new neuroprotective agents.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings

Patients with ocular hypertension

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings except presence of ocular hypertension (defined as untreated IOP ≥ 21 mmHg on at least three measurements in the medical history, no signs of glaucomatous damage in the optic disc or the glaucoma hemifield test)

Patients with primary open angle glaucoma

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Diagnosis of manifest primary open angle glaucoma (defined as pathological optic disc appearance, glaucoma hemifield test outside normal limits and untreated IOP > 20 mmHg on at least three measurements in the medical history)
* Mean Deviation in the visual field test ≥ 10dB

Patients with normal-tension glaucoma

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Diagnosis of normal-tension glaucoma (defined as pathological optic disc appearance, glaucoma hemifield test outside normal limits and untreated IOP ≤ 20 mmHg on at least three measurements in the medical history)
* Mean Deviation in the visual field test ≥ 10dB

Exclusion Criteria:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Exfoliation glaucoma, pigmentary glaucoma, history of acute angle closure
* Intraocular surgery within the last 6 months
* Ocular inflammation or infection within the last 3 months
* Pregnancy, planned pregnancy or lactating
* Any metallic, electric, electronic or magnetic device or object not removable except dental fillings
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
High resolution functional and structural imaging of the visual pathway | once on the study day (approximately 1 hour)
  The visual pathway will be imaged with 7-Tesla MRI. The images will be compared between the study groups.

SECONDARY OUTCOMES:
Retinal nerve fiber thickness | once on the study day (approximately 10 minutes)
  Parameters obtained from GDX and OCT measurements will be compared between groups.
Visual field test | once on the study day (approximately 20 minutes)
  Parameters from the Humphrey visual field test will be used for classification of severity of glaucoma or to prove that subjects are healthy.
Intraocular Pressure | once on the study day (1 minute)
  Goldmann applanation tonometry will be used for measurement of intraocular pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria